CLINICAL TRIAL: NCT04482829
Title: Efficacy and Safety of Jing-yuan-kang Granule in the Treatment of Lung Adenocarcinoma
Brief Title: TCM in the Treatment of Lung Adenocarcinoma
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: Henan University of Traditional Chinese Medicine (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: TCM for lung adenocarcinoma
Record Dates: First submitted 2020-07-03; First posted 2020-07-23 (Actual); Last update posted 2020-07-23 (Actual); Status verified 2020-07

CONDITIONS: Lung Adenocarcinoma
MeSH Terms: conditions — Adenocarcinoma of Lung

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Experimental Group (Experimental): On the basis of PC chemotherapy and symptomatic treatment, the patients in the experimental group will receive jing-yuan-kang granule with one dose daily.
  Interventions: Drug: Jing-yan-kang Granule; Drug: PC chemotherapy and symptomatic treatment
- Control Group (Other): All the patients in control group will receive PC chemotherapy and symptomatic treatment without other treatment.
  Interventions: Drug: PC chemotherapy and symptomatic treatment

INTERVENTIONS:
Drug: Jing-yan-kang Granule — Jing-yuan-kang granule will be administered 6 days on and 1 days off for 12weeks.
  Arms: Experimental Group
Drug: PC chemotherapy and symptomatic treatment — Drugs used in PC chemotherapy includes Pemetrexed and Cisplatin. Pemetrexed disodium for injection 500 mg per square meter, intravenous drip on day 1 in each treatment cycle.
  Cisplatin injection 75 mg per square meter, intravenous drip from day 1 to day 3 in each treatment cycle. One treatment cycle will be continued for 21 days and 4 cycles will be performed.
  If necessary, symptomatic treatment will also be used.

SUMMARY:
This study is to evaluate the efficacy and safety of Jin-yuan-kang granule in the treatment of lung adenocarcinoma (LUAD) preliminarily, and provide reference for further study.

DETAILED DESCRIPTION:
Lung adenocarcinoma (LUAD) is a type of non-small cell lung cancer (NSCLC) with a rapid disease progression and poor treatment effect. The LUAD patients have a short median survival time with 8-11 months. Up to now, chemotherapy is still the first-line treatment for LUAD. PC protocol (pemetrexed + cisplatin) is most commonly used, which is also recommended by NCCN guidelines. However, critical side effects have limited the application and efficacy. Patients will undergo poor quality of life, and the disease will progress rapidly. We still face the stern situation for the treatment of LUAD. It is urgent to develop new treatment and management strategies. Our previous study showed that jing-yuan-kang granule has certain curative effect on LUAD.

This is a multi-certers, randomized, controlled clinical trial to assess the efficacy and safety of Jing-yuan-kang granule in improving quality of life for LUAD patients. After a 2-week wash-out period, a total of 144 LUAD patients will be randomly assigned into experimental or control group with a ratio of 1:1. On the basis of that all the participants will receive PC chemotherapy and symptomatic treatment, the patients in the experimental group will receive jing-yuan-kang granule with no other treatments for control group. The primary outcome is quality of life. The secondary outcomes include Karnofsky (KPS) scores, clinical symptoms, and change of tumor volume. Safety and adverse events will also be assessed.

ELIGIBILITY:
Inclusion Criteria:

* A confirmed diagnosis of LADC.
* Age ranges from17years to75years.
* A KPS score ≥40.
* Without radiotherapy, immunotherapy and targeted therapy.
* Without participanting in any other trial.
* With signed informed consent.

Exclusion Criteria:

* Pregnant, nursing or may become pregnant women.
* The patient has a history of allergy to any of the components of the intervention drug;
* Patients with severe liver and kidney dysfunction, cardiovascular and cerebrovascular diseases.
* Unconscious or unable to communicate normally.
* Patients with poor compliance.

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 144 (Estimated)
Dates: Start 2020-09-15 (Estimated); Primary Completion 2020-12-30 (Estimated); Study Completion 2022-06-30 (Estimated)

PRIMARY OUTCOMES:
The quality of life will be evaluated by The European Organization for Research and Treatment of Cancer Quality of life Questinnaire Core-30(EORTC QLQ-C30) scale | Change at 3 weeks, 6 weeks, 9 weeks, and 12 weeks after treatment compared to baseline.
  A score of 1-4 will be administrated for each item in EORTC QLQ-C30 . The higher scores will indicate the worse outcomes.
Quality of life will be evaluated by Quality of life Questinnaire Lung Cancer-13(QLQ-LC13) | Change at 3 weeks, 6 weeks, 9 weeks, and 12 weeks after treatment compared to baseline.
  A score of 1-4 will be administrated for each item in QLQ-LC13. The higher scores will indicate the worse outcomes.

SECONDARY OUTCOMES:
Karnofsky(KPS) scores | Change at 3 weeks, 6 weeks, 9 weeks, and 12 weeks after treatment compared to baseline.
  Physical conditions will be evaluated by KPS scores with a score of 0-100. A higher score will indicate a better physical conditon.
TCM syndrome index | Change at 3 weeks, 6 weeks, 9 weeks, and 12 weeks after treatment compared to baseline.
  TCM symptom index will be recorded and calculated referring to the Guiding Principles of Clinical Research of New Chinese Medicine Treating Primary Bronchial Lung Cancer (2002 Edition) published by National Medical Products Administration of China. A total of scores of all the related symptoms will be calculated with a 0-4 for each symptom at baseline and after treatment. A higher value will indicate a worse symptom. The difference of TCM symptoms between baseline and posttreatment will be calculated first. Then, we will obtain the TCM syndrome index by the ratio between the above difference and the scores at baseline.
Change of tumor volume | Change at 12 weeks after treatment compared to baseline.
  Change of tumor volume will be assessed by the length of longest diameter. The longger diameter will indicate worse disease.
Adverse events will be evaluated and recorded at any time. | at baseline, up to 6 weeks and 12 weeks after treatment.
  Safety